CLINICAL TRIAL: NCT05687539
Title: The Effect of Mastiha Products on Functional Dyspepsia. A Randomised Crossover Study.
Brief Title: Mastiha or Mastiha Water in Functional Dyspepsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, Andriana C. Kaliora, Professor, Harokopio University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MASTIHA-WATER-FD
Record Dates: First submitted 2022-11-28; First posted 2023-01-18 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Functional Dyspepsia
MeSH Terms: interventions — mastiha

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Mastiha water (Experimental): Patients will receive 10ml of Mastiha water before every meal for one month
  Interventions: Dietary Supplement: Mastiha water
- Mastiha capsules (Experimental): Patients will receive 2 Mastiha capsules (2x350mg) before every meal for one month
  Interventions: Dietary Supplement: Mastiha capsules
- Control-Mastiha free (No Intervention): Patients will follow a Mastiha free one month period

INTERVENTIONS:
Dietary Supplement: Mastiha water — 10ml of mastiha water before every meal for one month
  Arms: Mastiha water
Dietary Supplement: Mastiha capsules — 2x350mg mastiha capsules before every meal for one month
  Arms: Mastiha capsules

SUMMARY:
The main aim of this study is to establish whether Mastiha products ameliorate functional dyspepsia symptoms.

DETAILED DESCRIPTION:
Functional dyspepsia has an approximate prevalence of 20% and is one of the main causes of upper abdominal discomfort. Its pathogenesis remain unclear and therapeutic options remain limited with patients seeking alternative therapies in herbal remedies. Mastiha has been proven to significantly improve symptoms in patients with functional dyspepsia compared to placebo. In the present study, the investigators aim to determine whether Mastiha capsules or Mastiha water have a better effect on the improvement of functional dyspepsia symptoms. Therefore, the investigators designed a randomized, three-way cross-over clinical trial. Fifty patients with functional dyspepsia, will be randomized over three treatment sequences of 30 days each, separated by 14-day washout periods. The three treatments will be: Mastiha capsules, Mastiha water or Mastiha free treatment. The primary outcome, which will be assessed by intention to treat, will be the Leuven Postprandial Distress Scale, a validated instrument for the assessment of symptoms in functional dyspepsia, supported by the European Medicines Agency.

ELIGIBILITY:
Inclusion Criteria:

functional dyspepsia diagnosis according to

* Rome criteria
* negative urea breath test for Helicobacter pylori
* upper gastrointestinal tract endoscopy with biopsy

Exclusion Criteria:

* organic diseases, such as peptic ulcer, gastrointestinal neoplasms, gastroesophageal reflux, irritable bowel syndrome
* pregnancy or lactation
* history of abdominal surgery or actinotherapy
* mental illness
* Severe impairment of heart, liver, or kidney function or respiratory function
* Alcohol overuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in Leuven Postprandial Distress Scale (LPDS) | 1 month
  The change in Leuven Postprandial Distress Scale will be evaluated at follow-up. LPDS minimum score is 0 and maximum 32. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change in quality of life | 1 month
  Change in quality of life at follow-up as assessed via the EQ-5D-5L questionnaire. EQ-5D-5L has a scale from 0 to 100, with higher scores meaning better outcomes.
Use of medicines | 1 month
  The percentage of patients that changed drug dose of medicines for functional dyspepsia will be evaluated at follow-up.
Change in anxiety | 1 month
  Change in anxiety at follow-up as assessed via the GAD-7 ANXIETY questionnaire. GAD-7 ANXIETY has a scale from 0 to 21, with higher scores meaning worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Andriana C. Kaliora, Ass. Prof., Study Director — Harokopio University
Locations (1):
- Andriana Kaliora, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kleftaki SA, Amerikanou C, Tzavara C, Biagki T, Sigala D, Bouziou A, Zouboulaki S, Koutsia A, Smyrnioudis EV, Anapliotis P, Kaliora AC. A randomized, three-way crossover clinical trial on the efficacy of Mastiha based therapies (Pistacia lentiscus var. Chia) in functional dyspepsia. Pharmacol Res. 2025 Dec;222:108019. doi: 10.1016/j.phrs.2025.108019. Epub 2025 Nov 4. PMID 41197785